CLINICAL TRIAL: NCT05677503
Title: Determination of the Relationship Between Red Cell Distribution Width, NT-proBNP and cTnT in Acute Myocardial Infarction Patients
Brief Title: Determination of the Red Cell Distribution Width, NT-proBNP and cTnT in Acute Myocardial Infarction Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hemat Kamel Maarouf, Resident doctor at clinical and chemical pathology department, Sohag University
Other Study IDs: Sohag_Med_22_12_07
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC — measurement of CBC will be performed at the time of admission and by the time of discharge
Diagnostic Test: (NT-proBNP) — measurement of serum NT-proBNP levels will be performed at the time of admission and by the time of discharge
Diagnostic Test: (cTnT) — measurement of cTnT levels will be performed at the time of admission and by the time of discharge

SUMMARY:
the study is to investigate the relationship of several parameters of complete blood count (CBC) including RDW with N-terminal pro-B-type natriuretic peptide (NT-proBNP) and cardiac troponin T (cTnT) in a cohort of acute myocardial infarction (AMI) patients.

DETAILED DESCRIPTION:
Patients and methods:

* Type of study: Observational prospective study
* Place of study: Sohag cardiology and gastroenterology center, department of cardiology and cardiac care unit.
* Ethical considerations: This research will be revised by the Scientific Ethical Committee of Sohag University Hospital. Consents will be taken from all patients.
* Study Methods:

  * A prospective study on 30 patients diagnosed as acute myocardial infarction on which measurement of CBC, serum NT-proBNP, and cTnT levels will be performed at the time of admission and by the time of discharge.

    1. Full history:

       1. Personal history: e.g. age, sex and smoking.
       2. Family history of cardiac diseases
       3. Medical history of: Hypertension, Ischemic heart disease, prior coronary artery bypass grafting, Prior Percutaneous coronary intervention, Prior Stroke, Prior Atrial fibrillation, therapeutic history
    2. Detailed clinical examination
    3. Electrocardiogram
    4. Laboratory investigation:

       1. Routine investigation in the form of CBC including RDW
       2. Specific investigation which include NT-proBNP and cTnT

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as acute myocardial infarction

Exclusion Criteria:

Patient with

* Decompensated heart failure
* Pulmonary hypertention
* Acute pulmonary embolism
* Septic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: _All patients included in the study will be subjected to:
  1. Full history:
     1. Personal history: e.g. age, sex and smoking.
     2. Family history of cardiac diseases
     3. Medical history of: Hypertension, Ischemic heart disease, prior coronary artery bypass grafting, Prior Percutaneous coronary intervention, Prior Stroke, Prior Atrial fibrillation, therapeutic history
  2. Detailed clinical examination
  3. Electrocardiogram
  4. Laboratory investigation:
     1. Routine investigation in the form of CBC including RDW
     2. Specific investigation which include NT-proBNP and cTnT
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
complete blood count (CBC) | 7 months
  measurement of CBC levels will be performed
Level of (NT-proBNP) | 7 months
  measurement of serum NT-proBNP level will be performed
Level of (cTnT) | 7 months
  measurement of cTnT level will be performed